CLINICAL TRIAL: NCT03646422
Title: Spanish Academy of Dermatology and Venereology (AEDV) Registry of Primary Cutaneous Lymphoma
Brief Title: AEDV Registry of Primary Cutaneous Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Academia Española de Dermatología (Other)
Responsible Party: Sponsor
Other Study IDs: FAE-LIN-2016-01
Record Dates: First submitted 2018-07-18; First posted 2018-08-24 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Lymphoma, T-Cell, Cutaneous; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse; Sezary Syndrome; Lymphoma, Extranodal NK-T-Cell; Lymphoma, B-Cell
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse; Sezary Syndrome; Lymphoma, Extranodal NK-T-Cell; Lymphoma, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Registry of patients (exposure is Cutaneous Lymphoma)

SUMMARY:
Registry of patients with Primary Cutaneous Lymphoma seen at participating centers in Spain. The registry will identify patients with this disease and includes information about stage, diagnostic and therapeutic interventions and willingness to participate in further studies.

DETAILED DESCRIPTION:
Registry of patients with Primary Cutaneous Lymphoma seen at participating centers in Spain. The registry will identify patients with this disease and includes information about stage, diagnostic and therapeutic interventions and willingness to participate in further studies.

Data is entered in the registry in each of the participating cutaneous lymphoma clinics. These data are updated at least yearly. Participants receive specific training before starting, and there is an online continuous monitoring system.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with primary cutaneous lymphoma

Exclusion Criteria:

* Not willing to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population should be an accurate representation of patients with primary cutaneous lymphoma in Spain
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Maximum TNM stage | Through study completion, an average every 1 year
  Proportion
Therapeutic groups used | Through study completion, an average every 1 year
  Including drugs, phototherapy, radiotherapy and procedures (blood marrow transplant)
Mortality | Through study completion, an average every 1 year
  Rate

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Ortiz, MD, PhD, Principal Investigator — Hospital 12 de Octubre
Locations (14):
- Spain (14):
  - Hospital Clinic, Barcelona
  - Hospital Universitario Basurto, Bilbao
  - Hospital General de Ciudad Real, Ciudad Real
  - hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - C.H.U. Insular-Materno Infantil, Las Palmas de Gran Canaria
  - H.U. Fundación Jiménez Díaz, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario Príncipe de Asturias, Madrid
  - Complejo Hospitalario de Navarra, Pamplona
  - CHOP-Hospital de Montecelo, Pontevedra
  - H.U. Nuestra Señora de la Candelaria, Santa Cruz de Tenerife
  - H.U. Virgen del Rocío, Seville
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Valencia-Clínico Malva-Rosa, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Penate Y, Servitje O, Machan S, Fernandez-de-Misa R, Estrach MT, Acebo E, Mitxelena J, Ramon MD, Florez A, Blanes M, Morillo M, Medina S, Bassas J, Zayas A, Espinosa P, Perez A, Gonzalez-Romero N, Dominguez JD, Muniesa C, Lopez Robles J, Combalia A, Yanguas I, Suh H, Polo-Rodriguez I, Bielsa I, Mateu A, Ferrer B, Descalzo MA, Garcia-Doval I, Ortiz-Romero PL. The First Year of the AEVD Primary Cutaneous Lymphoma Registry. Actas Dermosifiliogr (Engl Ed). 2018 Sep;109(7):610-616. doi: 10.1016/j.ad.2018.03.006. Epub 2018 Apr 19. English, Spanish. PMID 29680323